CLINICAL TRIAL: NCT04044651
Title: A Randomized, Phase IIb Study of Lenvatinib Plus Nivolumab Versus Lenvatinib for Advanced Hepatocellular Carcinoma (HCC) With Hepatitis B Virus (HBV) Infection
Brief Title: Lenvatinib Plus Nivolumab Versus Lenvatinib for Advanced Hepatocellular Carcinoma With Hepatitis B Virus Infection
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Bristol-Myers Squibb company terminated this study
Sponsor: Shi Ming (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Guangzhou No.12 People's Hospital (Other Government); Guangdong Provincial People's Hospital (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor-Investigator, Shi Ming, Proffessor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC-S051
Record Dates: First submitted 2019-07-31; First posted 2019-08-05 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Lenvatinib; Nivolumab; Hepatitis B virus
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis B | interventions — lenvatinib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lenvatinib plus nivolumab (Experimental): nivolumab 480 mg IV infusions for 30 minutes q4w+ lenvatinib 12 mg (or 8 mg) by mouth (Po) once daily
  Interventions: Drug: Lenvatinib; Drug: Nivolumab
- Lenvatinib (Active Comparator): Lenvatinib 12 mg (or 8 mg) Po once daily
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib — lenvatinib 12 mg (or 8 mg) by mouth (Po) once daily
  Other Names: E7080, Lenvima
Drug: Nivolumab — nivolumab 480 mg IV infusions for 30 minutes q4w
  Arms: Lenvatinib plus nivolumab

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of lenvatinib plus nivolumab compared with lenvatinib monotherapy for patients with advanced hepatitis B virus infection-related hepatocellular carcinoma.

DETAILED DESCRIPTION:
Lenvatinib was non-inferior to sorafenib in overall survival in untreated advanced hepatocellular carcinoma, and nivolumab was effective and tolerable in patients with advanced hepatocellular carcinoma. No study has evaluated the efficacy and safety of lenvatinib plus nivolumab compared with lenvatinib monotherapy. Thus, the investigators carried out this prospective, randomized, phase IIb study to find out it.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all of the following criteria in screening tests and observations within 14 days before enrollment will be included in the study.

1. Signed Informed Consent Form
2. Males and Females, 18 years or older at time of signing Informed Consent Form
3. Ability to comply with the study protocol, in the investigator's judgment
4. HCC with diagnosis confirmed by histology/cytology by AASLD criteria
5. Barcelona clinic liver cancer (BCLC) C stage.
6. No prior systemic therapy for HCC
7. Patients must not be appropriate for surgery or loco-regional therapy. Patients can receive no previous anti-cancer therapy or have progressed or have intolerable adverse events after surgery or loco-regional therapy. Surgery or locoregional therapy include hepatic resection, ablation, transcatheter arterial chemoembolization (TACE), hepatic arterial infusion chemotherapy (HAIC), radiotherapy, and must have been completed at least 4 weeks (washout period) prior to the baseline scan. In addition, all acute toxic effects of the locoregional procedure must have resolved to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 Grade<=1.
8. At least one tumor lesion that can be accurately measured according to the RECIST 1.1
9. ECOG Performance Status of 0 or 1
10. No cirrhosis or cirrhotic status of Child-Pugh class A only. Documented virology status of HBV, as confirmed by screening HBV serology test, as evidenced by detectable HBV surface antigen. (there is no lower and upper limit of HBV DNA, but patients must be on effective antiviral therapy if HBV DNA is positive [greater than zero]).
11. Adequate hematologic and end-organ function, defined by the following laboratory test results, obtained within 14 days prior torandomization, unless otherwise specified:

    1. white blood cell count ≥ 3.0×10⁹ per L
    2. absolute neutrophil count ≥ 1.5×10⁹ per L
    3. platelet count ≥ 75×10⁹ per L
    4. Hemoglobin ≥ 8.5 g/dL
    5. Prothrombin time (PT)-international normalized ratio (INR) ≤ 2.3 or Prothrombin time (PT) ≤ 6 seconds above control
    6. total bilirubin ≤ 30mmol/L
    7. serum albumin ≥ 30 g/L
    8. aspartate transaminase and alanine transaminase ≤ 5×upper limit of the normal
    9. creatinine clearance of ≤1.5×upper limit of the normal or a creatinine clearance > 50 mL/min (Cockcroft-Gault formula)
    10. left ventricular ejection fraction (LEVF) ≥45% as measured by echocardiography
12. Reproductive status: Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within one day prior to the start of study drug. Women must not be breastfeeding.

Exclusion Criteria:

Patients who meet one of the following criteria in screening tests and observations before enrollment will be excluded from the study:

1. Fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC was excluded.
2. Any history of hepatic encephalopathy
3. Any prior (within 30 days) or current clinically significant gastrointestinal bleeding or clinically significant ascites as measured by physical examination and that requires active paracentesis for control
4. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
5. Known history of hepatitis C virus (HCV) or hepatitis D virus (HDV) infection
6. Active bacterial or fungal infections requiring systemic treatment within 7 days prior to study drug dosing
7. Prior organ allograft such as liver transplant, etc. or allogeneic bone marrow transplantation
8. Known or suspected allergy to the investigational agents or any agent given in association with this trial
9. Subjects with any active autoimmune disease or history of known or suspected autoimmune disease except for subjects with vitiligo, resolved childhood asthma/atopy, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement. psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
10. Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg/day prednisone equivalent) or other immunosuppressive medications within 30 days of study administration. Inhaled or topical steroids are permitted in the absence of active autoimmune disease
11. Treatment with anti-platelet therapy (aspirin at dose>=300 mg/day, clopidogrel at dose>=75 mg/day) or current anticoagulation therapy
12. Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody (or any other antibody or drug specifically targeting T-cell costimulation or checkpoint pathways)
13. All toxicities attributed to prior anti-cancer therapy other than neuropathy, alopecia and fatigue must have resolved to Grade 1 (NCI CTCAE version 4.03) or baseline before administration of study drug. Subjects with toxicities attributed to prior anti-cancer therapy which are not expected to resolve and result in long lasting sequelae are permitted to enroll. Neuropathy must have resolved to Grade 2 (NCI CTCAE version 4.03).
14. Known central nervous system tumors including metastatic brain disease
15. Patients who are pregnant or breastfeeding. Women with a positive pregnancy test at enrollment or prior to administration of study medication
16. Other invasive malignant diseases
17. Prisoners, or subjects who are compulsory detained
18. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-30 (Estimated); Primary Completion 2021-03-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 18 months
  OS is the length of time from the date of randomization until death from any cause. The date survival was last confirmed will be used to censor surviving patients. In the absence of confirmation of death, the survival time will be censored at the last date the patient was known to be alive or at the cutoff date, whichever comes first. Unfollowable patients will be censored by the date survival was last confirmed before they became unfollowable.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 18 months
  ORR, as determined based on tumor response according to RECIST 1.1, is defined as the proportion of all randomized subjects whose best overall response (BOR) is either a CR or PR. BOR is determined by the best response designation recorded between the date of randomization and the date of first objectively documented progression or the date of subsequent anti-cancer therapy, whichever occurs first. For subjects without documented progression or subsequent anti-cancer therapy, all available response designations will contribute to the BOR determination. For a BOR of CR or PR, the initial response assessment must be confirmed by a consecutive assessment no less than 4 weeks (28 days) later.
Progression free survival (PFS) | 18 months
  PFS will be determined from assessments based on RECIST 1.1. PFS is defined as the time from the date of randomization to the date of the first objectively documented tumor progression or death due to any cause. Subjects who die without a reported prior progression and without initiation of subsequent anti-cancer therapy will be considered to have progressed on the date of their death. Subjects who did not progress or die will be censored on the date of their last tumor assessment. Subjects who did not have baseline tumor assessment will be censored on the date they were randomized. Subjects who did not have any on-study tumor assessments and did not die will be censored on the date they were randomized. Subjects who started any subsequent anti-cancer therapy without a prior reported progression will be censored at the last tumor assessment prior to subsequent anti-cancer therapy.
Duration of response (DOR) | 18 months
  DOR will be determined based on RECIST 1.1. DOR is time from documentation of tumor response to disease progression. Disease progression as assessed according to RECIST 1.1.
Adverse event | 18 months
  Safety will be evaluated according to the NCI CTCAE Version 4.03. All observations pertinent to the safety of the study medication will be recorded on the CRF and included in the final report. All adverse events, whether considered treatment-related or not, will be reported on the CRF with diagnosis, start/stop dates, action taken, whether treatment was discontinued, any corrective measures taken, outcome and other possible causes.
OS stratified according to degree of PVTT (Vp0-3 vs Vp4) | 18 months
  To compare the OS of nivolumab plus lenvatinib to lenvatinib stratified according to degree of PVTT (Vp0-3 vs Vp4)

OTHER OUTCOMES:
Disease control rate (DCR) | 18 months
  DCR will be determined based on RECIST 1.1. DCR is defined as the rate of complete response (CR) plus partial response (PR) plus stable disease (SD). Tumor response includes assessment of target lesions, nontarget lesions and new lesions. CR and PR will be confirmed at least 4 weeks after the first observation.
Time to progression (TTP) | 18 months
  TTP was defined as the time from the date of randomization to the date of first documentation of disease progression based on RECIST 1.1.
Time to response (TTR) | 18 months
  TTR is time from the date of randomization to the date of tumor response.
Rates and degrees of HBV DNA breakthrough | 18 months
  To evaluate rates and degrees of HBV DNA breakthrough of patients that receive nivolumab plus lenvatinib and patients that receive lenvatinib. HBV DNA breakthrough is that HBV-infected patients had >1 log increase in HBV DNA.
Cancer-related QoL | 18 months
  To assess the subject's cancer-related QoL using the Functional Assessment of Cancer Therapy-Hepatobiliary (FACT-Hep) questionnaire
Surgical conversion rate | 18 months
  To assess surgical conversion rate of patients that receive nivolumab plus lenvatinib and patients that receive lenvatinib. Surgical conversion rate is that incidence rate of patients that receive surgical resection.
PD-L1 biomarker | 18 months
  To assess the PD-L1 biomarker of patients that receive nivolumab plus lenvatinib and patients that receive lenvatinib.
OS stratified according to presence or absence of extrahepatic metastasis, HBV DNA level, AFP level, or ECOG score | 18 months
  To compare the OS of nivolumab plus lenvatinib to lenvatinib stratified according to presence or absence of extrahepatic metastasis, HBV DNA level (no more than 500 IU/ml vs more than 500 IU/ml), AFP level (no more than 400 ng/ml vs more than 400 ng/ml), or ECOG score (0 vs 1), respectively.
AFP level change | 18 months
  To asess AFP level change of patients that receive nivolumab plus lenvatinib and patients that receive lenvatinib.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Shi, MD, Principal Investigator — Sun Yat-sen University
Locations (5):
- China (5):
  - Cancer Center Sun Yat-sen University, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Third Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Guangzhou Twelfth People 's Hospita, Guangzhou, Guangdong